CLINICAL TRIAL: NCT07355348
Title: Codesign of a Cognitive Stepped Care Program (CSCP) to Enhance Quality of Life in Adults With Brain Metastases: Evaluation of Feasibility, Acceptability and Preliminary Efficacy
Brief Title: Feasibility of a Cognitive Stepped Care Program for Adults With Brain Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Samantha Mayo, Clinician Investigator, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-5444.0
Record Dates: First submitted 2025-12-31; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Brain Metastases; Brain Metastasis
Keywords: cancer-related cognitive impairment; brain metastases; brain metastasis; stepped care; symptom management
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Stepped Care Program (Experimental)
  Interventions: Behavioral: Cognitive Stepped Care Program (CSCP)

INTERVENTIONS:
Behavioral: Cognitive Stepped Care Program (CSCP) — The Cognitive Stepped Care Program comprises two steps:
  1. Cognitive Symptom Screening: Patients will complete a 10-item cognitive screening tool. Each item is rated from 0-10, with thresholds for mild, moderate and severe symptoms.
  2. Cognitive Symptom Management. Patients will receive a cognitive symptom management intervention tailored to their symptom severity. Symptom management interventions will be based on the highest response score across the 10-item screening tool, ranging from no support (no symptoms), to educational materials (mild symptoms), to computerized cognitive testing with an individualized debrief (moderate-severe symptoms), with group strategy training and/or neuropsychological consultation provided as needed.

SUMMARY:
Background: Cognitive symptoms are common and often severe in patients with brain metastases, significantly impacting their quality of life and ability to manage cancer care. Currently, there is no standard approach for routinely assessing and managing these symptoms in oncology clinics.

Objective: This study aims to evaluate the feasibility, acceptability, and preliminary efficacy of the Cognitive Stepped Care Program (CSCP) in a Brain Metastases Clinic.

Methods: This is a prospective, mixed-methods feasibility study involving patients with brain metastases, their caregivers, and clinic staff. Patients will undergo routine cognitive symptom screening using a standardized tool. Based on symptom severity, they will receive tiered interventions ranging from no support, to education materials, to computerized cognitive testing with individualized debrief, with group strategy training and/or neuropsychological consultation, as needed. Patients will complete questionnaires before and after the intervention regarding their symptoms and quality of life. Patients, caregivers and staff will provide their feedback about the intervention through questionnaires and interviews.

Outcomes: Primary outcomes include feasibility and acceptability of the CSCP. Secondary outcomes include preliminary changes in cognitive symptoms, self-efficacy, and quality of life.

Significance: This study will inform the potential integration of a structured cognitive support program into standard care for patients with brain metastases and may provide a model for similar interventions in other oncology settings.

ELIGIBILITY:
Patients:

Inclusion Criteria:

* Diagnosed with a brain metastasis for any primary cancer
* Receiving follow-up care in the Brain Metastases Clinic
* Adult (≥ 18 years)
* Able to speak, read, and write in English
* Able to provide written informed consent

Exclusion Criteria:

* History of significant developmental/learning disability or psychiatric disorder, acquired neurological disorder (e.g., traumatic brain injury)
* Poor performance status (ECOG ≥ 3)
* Life expectancy < 3 months

Caregivers:

Inclusion Criteria:

* Self-identified or identified by consenting patient as a primary caregiver for a person with brain metastases receiving follow-up in the Brain Metastases Clinic
* Adult (≥ 18 years)
* Able to speak, read, and write in English
* Able to provide written informed consent

Exclusion Criteria:

• N/A

Staff:

Inclusion Criteria:

* Currently working as a clinician or administrative staff member in the Brain Metastases Clinic
* Adult (≥ 18 years)
* Able to speak, read, and write in English
* Able to provide written informed consent

Exclusion Criteria:

• N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Intervention Completion Rate | Through study completion, an average of 1 month
  Proportion of patients who are able to complete the CSCP (i.e. complete the cognitive symptom management intervention as allocated to them based on cognitive screening score)
Intervention Satisfaction | Through study completion, an average of 1 month
  Rating on a 5-point Likert scale (0-poor to 4-excellent), with optional open-text item for additional comments
Descriptions of Feasibility | Through study completion, an average of 1 month
  Post-intervention qualitative interviews with participants (patients/caregivers one week after their last interaction of the CSCP, or staff at the completion of the study period) will also explore their perceptions of the feasibility and acceptability of the CSCP, including suggestions for improvement of the intervention.
Recruitment Rate | Baseline
  Proportion of eligible participants who are enrolled in the study
Retention Rate | Through study completion, an average of 1 month
  Proportion of patients who complete the study (i.e. pre-post data collection)

SECONDARY OUTCOMES:
Intervention Reach | Baseline
  We will examine the representativeness of the patients were enrolled in the CSCP. For all consented patient participants, we will collect demographic and clinical information through a study-specific questionnaire and a review of health records. This will be compared to historical patient demographics from the study setting.
Intervention Efficacy (Preliminary) - Change in Cognitive Symptom Severity | Baseline and up to 4 months
  Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog3)
Intervention Effectiveness (Preliminary) - Change in Perceived Self-Efficacy | Baseline and up to 4 months
  Patient-Reported Outcomes Measurement Information System - General Self-Efficacy (PROMIS 4-item General Self-Efficacy)
Intervention Effectiveness (Preliminary) - Change in Cancer-related Quality of Life | Baseline and up to 4 months
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC QLQ-C30)
Intervention Efficacy (Preliminary) - Change in Cancer-related Quality of Life - Brain-specific | Baseline and up to 4 months
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire BN-20 (EORTC QLQ-BN20) for brain-specific symptoms
Intervention Efficacy (Preliminary) - Perceptions | Up to 4 months
  Post-intervention qualitative interviews will include questions about what participants found most valuable (patients, caregivers, staff), the impact on their overall well-being (patients), and if there were, any negative experience associated with the CSCP (patients, caregivers, staff).
Intervention Adoption | Up to 1 year
  Post-intervention qualitative interviews will explore perceptions from patients, caregivers, and staff about the potential motivations for the adoption of the CSCP within the Brain Metastasis clinic and/or the organization more broadly. Questions will also gauge facilitators and barriers to this adoption.
Intervention Implementation - Factors Influencing CSCP Fidelity | Up to 1 year
  From CSCP case logs, we will collect the time spent per patient on the CSCP, any adverse events, and any challenges to implementation fidelity (e.g., scheduling, technical issues).
Intervention Implementation - Perceptions | Up to 1 year
  Interviews with patients, caregivers, and staff will gather feedback on challenges to implementation and what strategies, tools, or infrastructure would need to be developed to better ensure that the intervention is delivered as intended.
Intervention Maintenance | Up to 1 year
  Staff interviews will explore anticipated facilitators and barriers to long-term implementation within standard care, including its impact on other services.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Not currently included in the approved protocol